CLINICAL TRIAL: NCT03245190
Title: Efficacy and Safety of Chiauranib in Advanced Hepatocellular Carcinoma: a Single-arm, Open-label, Multi-center, Exploratory Phase Ib Study
Brief Title: Study of Chiauranib in Patients With Advanced Hepatocellular Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chipscreen Biosciences, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAR104
Record Dates: First submitted 2017-08-04; First posted 2017-08-10 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — chiauranib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chiauranib (Experimental): Patients take Chiauranib capsules 50mg, orally once daily, 28 days as a cycle.
  Interventions: Drug: Chiauranib

INTERVENTIONS:
Drug: Chiauranib — 50mg, orally once daily
  Other Names: CS2164

SUMMARY:
Chiauranib, which simultaneously targets against VEGFR/Aurora B/CSF-1R, several key kinases involved in tumor angiogenesis, tumor cell mitosis, and chronic inflammatory microenvironment.

DETAILED DESCRIPTION:
Chiauranib is a novel orally active multi-target inhibitor that simultaneously inhibits the angiogenesis-related kinases (VEGFR2, VEGFR1, VEGFR3, PDGFRa and c-Kit), mitosis-related kinase Aurora B and chronic inflammation related kinase CSF-1R in a high potency manner with the IC50 at a single-digit nanomolar range. In particular, Chiauranib showed very high selectivity in the kinase inhibition profile with little activity on off-target non-receptor kinases, proteins, GPCR and ion channels, indicative of a better drug safety profile in terms of clinical relevance.

Because of its broad preclinical anti-tumor efficacy and the potential to improve conventional TKI kinase inhibitor therapy in various cancer indications, Chiauranib has now entered phase Ib clinical trials.

This clinical trial is studying the efficacy and safety of chiauranib works in treating patients with advanced hepatocellular carcinoma, in the meantime, exploring the latent biomarkers accompany with chiauranib, as well as the relevancy of which and clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age ≥ 18 years and ≤70 years.
2. Histological or cytological confirmation of HCC (hepatocellular carcinoma) or non-invasive diagnosis of HCC as per American Association for the Study of Liver Diseases criteria in patients with a confirmed diagnosis of cirrhosis.
3. Barcelona Clinic Liver Cancer stage Category B or C that cannot benefit from treatments of locoregional therapy, or provided that progression has been documented after these therapies.
4. Patients should have failed or been intolerant of at least one prior systemic therapy regimen which could include systemic chemotherapy (such as oxaliplatin, arsenious acid) and/or sorafenib.
5. At least one uni-dimensional measurable lesion according to RECIST (RECIST version 1.1), and modified RECIST for HCC (mRECIST)：a. HCC lesions should have at least one accurate repeated dimension as 1 cm or more ); b. extrahepatic lesions: a lymph node must be 1.5 cm or more in short axis, and Non-lymph node lesions must be at least 1 cm in longest diameter. Tumor lesions situated in a previously irradiated area, or in an area subjected to other loco-regional therapy, may be considered measurable if there has been demonstrated progression in the lesion.
6. Liver function status Child-Pugh Classification with score ≤ 7 points. Child Pugh status should be calculated based on clinical findings and laboratory results during the screening period.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
8. Laboratory criteria are as follows (laboratory results within 7 days prior to first dose, and without receiving any supportive treatment for the following parameters within 2 weeks from the last dose prior to study entry):

   1. Complete blood count: white blood cell count ≥ 3.0×109/L; absolute neutrophil count (ANC) ≥1.5×109/L ;hemoglobin (Hb) ≥85g/L ; platelets >=60×109/L
   2. Biochemistry test: total bilirubin≦1.5×ULN; alanine aminotransferase(ALT) ,aspartate aminotransferase(AST)≦5×ULN ; plasma albumin≥ 28 g/L; serum creatinine(cr)≦1.5×ULN; serum amylase≦1.5×ULN;
   3. Coagulation test: International Normalized Ratio (INR) < 1.5; activated partial thromboplastin time (APTT) < 1.5×ULN
   4. Thyroid function test: thyroid stimulating hormone (TSH) < 10mIU/L；
9. Life expectancy of at least 12 weeks.
10. All patients must have given signed, informed consent prior to registration on study.

Exclusion Criteria:

1. Any target treatment like sorafenib within 2 weeks prior to first dose of study drug; With the exception of target treatment, any anti-cancer systemic treatment (including chemotherapy, immunotherapy, radiotherapy, and anti-cancer Chinese traditional medicine, et al) or locoregional therapy (including but not limited to surgery, radiofrequency ablation or transarterial chemoembolization ) within 4 weeks prior to first dose of study drug; any supportive treatment for haematology (including transfusion, blood products, or drugs that stimulate blood cells growth like G-CSF, et al) within 2 weeks prior to first dose of study drug.
2. Known Cholangiocarcinoma or Fibrolamellar Hepatocellular Carcinoma; Known history of, or ongoing second primary cancer, except: adequately treated basal cell or squamous cell skin cancer, curatively treated in-situ cancer of the cervix, unless received curative treatment and with documented evidence of no recurrence during the past five years;
3. Known metastatic brain or meningeal tumors
4. Patients with uncontrolled or significant cardiovascular disease, including:

   1. Grade II or higher Congestive heart failure, unstable angina pectoris, myocardial infarction (NYHA Classification) within 6 months prior to study entry; or arrhythmia requiring treatment, or Left Ventricular Ejection Fraction (LVEF) < 50% during screening stage.
   2. Primary cardiomyopathy (dilated cardiomyopathy, hypertrophic cardiomyocyte, arrhythmogenic right ventricular cardiomyopathy, restrictive cardiomyopathy, et,al).
   3. History of significant QT interval prolongation, or Corrected QT Interval QTc≥450ms(male), QTc≥470ms（female）at screening.
   4. Symptomatic coronary heart disease requiring treatment.
   5. Uncontrolled hypertension (> 140/90 mmHg) with single medication.
5. History of active bleeding within 6 months or esophageal varices bleeding led by portal hypertension within 2 months prior to screening ; or patients receiving anticoagulation therapy; or patients with evidence of GI bleeding potential.
6. Uncontrolled ascites or pleural effusion (defined as not easily controlled with diuretic or paracentesis treatment).
7. History of transjugular intrahepatic portosystemic shunts (TIPSS).
8. History of abdominal fistula, gastrointestinal perforation or abdominal abscess within 28 days prior to screening.
9. History of deep vein thrombosis or pulmonary embolism.
10. History of interstitial lung disease(ILD), or with ongoing signs and symptoms at the time of screening.
11. History of hypothyroidism; or patients receiving substitutional treatment with thyroid hormone.
12. With any ongoing toxicities (>CTCAE grade 1) caused by previous cancer therapy.
13. Patients with factors that could affect oral medication (such as dysphagia, chronic diarrhea, intestinal obstruction etc), or undergone gastrectomy.
14. History of liver transplantation, or patients in preparation of liver transplantation.
15. 6 weeks or less from the last major surgery that involved general anaesthesia, or 2 weeks or less from the last minor surgery prior to screening (excluding placement of vascular access ) .
16. Proteinuria positive(≥1g/24h).
17. Patients with active or unable to control infections including human immunodeficiency virus (HIV), or other serious infectious diseases.
18. Patients with untreated active hepatitis B virus (HBV) (HBsAg positive and HBV DNA ≥ 2000 IU/mL) . But patients with controlled(treated) HBV fulfilling the following criteria can be eligible for the study: HBV DNA< 2000 IU/mL , or patients on anti-HBV suppression with HBV DNA< 2000 IU/mL before study enrollment.
19. Patients with untreated active hepatitis C virus.
20. Any mental or cognitive disorder, that would impair the ability to understand the informed consent document, or limit compliance with study requirements/treatment.
21. Any previous treatment with aurora kinase inhibitors.
22. Candidates with drug abuse.
23. Women of childbearing potential not willing to use and utilize an adequate method of contraception (such as intrauterine device, contraceptive and condom) throughout treatment and for at least 12 weeks after the last dose; pregnant or breastfeeding women; the result of urine pregnancy test was positive at screening; Man participants not willing to use and utilize an adequate method of contraception throughout treatment.
24. Any other condition which is inappropriate for the study according to investigators' judgment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-04-28 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
16 weeks progression-free rate (16W-PFR) | Up to a minimum 16 weeks after the last participant's first dose, or progression, or died, whichever came first

SECONDARY OUTCOMES:
Rate of Treatment-Related Adverse Events in Study Participants | Up to a minimum 20 weeks after the last participant's first dose, or progression, or 75% subjects died, whichever came first, assessed up to 24 months
  Safety evaluation as measured by adverse events (AE), vital signs，electrocardiograph(ECG) and abnormal laboratory results according to CTCAE V4.03
Time to progression(TTP) | Approximately 24 months
Objective response rate (ORR) | Approximately 24 months
  ORR is defined as the percentage of participants whose best overall response is either complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 and modified RECIST for HCC (mRECIST), respectively.
Disease-control rate (DCR) | Approximately 24 months
Duration of response (DOR) | Approximately 24 months
Progression-free survival (PFS) | Approximately 24 months
Overall survival (OS) | Approximately 24 months
6 months progression-free rate | At 6 months
6 months overall survival rate | At 6 months
12 months overall survival rate | At 12 months

OTHER OUTCOMES:
Median score of immunohistochemical expressed by Aurora B、CSF-1R and Myc protein. | Assessed up to 24 months
Screening characteristics of ctDNA measurement (single gene analysis). | Assessed up to 24 months
Screening characteristics of ctDNA measurement (multi-gene analysis). | Assessed up to 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided